CLINICAL TRIAL: NCT01454050
Title: PME/Master Study of the Lumax 740 ICD Family
Brief Title: Lumax 740 Master Study
Acronym: Lumax 740
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 55
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Safety and Efficacy of the Lumax 740 ICD Family
Keywords: ICD therapy; RV/LV Capture Control; Safety and Efficacy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to prove the safety and efficacy of the Lumax 740 ICD family. Primarily, the newly implemented RV/LV Capture Control algorithm is evaluated, which automatically measures the RV/LV threshold and subsequently adjusts the pacing output.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Standard indication for single, dual, or triple chamber ICD.

  * Legal capacity and ability to consent
  * Signed patient informed consent

In addition for HF-T devices:

* Bipolar LV-lead with a min. distance of 15 mm between tip and ring
* True bipolar RV lead

Exclusion Criteria:

* Standard contraindication for single, dual, or triple chamber ICD.

  * Age < 18 years
  * Pregnant or breast-feeding woman
  * Cardiac surgery planned within the next 6 months
  * Life expectancy of less than 6 months
  * Participating in any other clinical study of an investigational cardiac drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard ICD indication who are referred to the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of the automatic Capture Control feature | PHD, 1-, 3- and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Klein, Prof. Dr., Study Chair — Herz im Zentrum Hannover, Germany
Locations (1):
- Medical School Hannover, Hanover, Germany